CLINICAL TRIAL: NCT00002692
Title: A RANDOMISED TRIAL OF INTRAVENOUS VERSUS INTRAHEPATIC ARTERIAL 5-FU AND LEUCOVORIN FOR COLORECTAL LIVER METASTASES
Brief Title: Intravenous Compared With Intrahepatic Chemotherapy in Treating Patients With Colorectal Cancer Metastatic to the Liver
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Medical Research Council (Other Government)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000064434; MRC-CR05; EU-95032
Record Dates: First submitted 1999-11-01; First posted 2004-05-21 (Estimated); Last update posted 2013-12-19 (Estimated); Status verified 2007-05

CONDITIONS: Colorectal Cancer; Metastatic Cancer
Keywords: stage IV colon cancer; stage IV rectal cancer; recurrent colon cancer; recurrent rectal cancer; adenocarcinoma of the colon; adenocarcinoma of the rectum; liver metastases
MeSH Terms: conditions — Colorectal Neoplasms; Neoplasm Metastasis; Colonic Neoplasms; Rectal Neoplasms | interventions — Fluorouracil; Leucovorin

INTERVENTIONS:
Drug: fluorouracil
Drug: isolated perfusion
Drug: leucovorin calcium

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Randomized phase III trial to compare the effectiveness of intravenous infusion or intrahepatic infusion of fluorouracil and leucovorin in treating patients with colorectal cancer metastatic to the liver.

DETAILED DESCRIPTION:
OBJECTIVES: I. Compare the survival and response rates of patients with colorectal liver metastases treated with intravenous vs. intrahepatic arterial infusion of fluorouracil/leucovorin. II. Assess the effect of these 2 treatments on symptoms and quality of life of these patients.

OUTLINE: Randomized study. Patients randomized to Arm II should have a preoperative hepatic angiography; at laparotomy, an intrahepatic arterial catheter is fused into the gastroduodenal artery to establish an infusion of both lobes of the liver. Arm I: Single-Agent Chemotherapy with Drug Modulation. Fluorouracil, 5-FU, NSC-19893; with Leucovorin calcium, CF, NSC-3590. Intravenous infusion. Arm II: Single-Agent Chemotherapy with Drug Modulation. 5-FU; with CF. Intrahepatic arterial infusion.

PROJECTED ACCRUAL: 312 patients are expected to be randomized within 3-4 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS: Histologically confirmed adenocarcinoma of the colon or rectum with metastases confined to the liver and not amenable to surgery

PATIENT CHARACTERISTICS: Age: Any age Performance status: WHO 0-2 Life expectancy: More than 3 months Hematopoietic: WBC at least 3,000/mm3 Absolute neutrophil count at least 1,500/mm3 Platelet count at least 100,000/mm3 Hepatic: Bilirubin less than 3.5 mg/dL (50 micromoles/liter) Renal: Not specified Cardiovascular: No uncontrolled heart disease (e.g., congestive heart failure, angina) Other: No uncontrolled infection No other uncontrolled medical illness

PRIOR CONCURRENT THERAPY: No prior fluorouracil (5-FU) for advanced disease More than 6 months since adjuvant 5-FU (e.g., in AXIS or QUASAR studies)

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 312 (Estimated)
Dates: Start 1994-12

CONTACTS AND LOCATIONS:
Overall Officials: David J. Kerr, MD, FRCP, DSc, Study Chair — University Hospital Birmingham
Locations (1):
- University Birmingham, Birmingham, England, United Kingdom

REFERENCES:
- [Result] McArdle C: IV versus IHA 5FU/leucovorin for colorectal liver metastases: preliminary results of the MRC CR05 EORTC 40972 randomised trial. [Abstract] Br J Cancer 85 (suppl 1): A-CT2. 1, 2001.
- [Result] McArdle C, Kerr DJ, Ledermann J, et al.: Intravenous (IV) vs intrahepatic (IHA) 5FU/leucovorin for colorectal (CRC) liver metastases: preliminary results of the MRC CR05/EORTC 40972 randomised trial. [Abstract] Proceedings of the American Society of Clinical Oncology 20: A-499, 2001.
- [Result] McArdle C, Kerr DJ, Ledermann J, et al.: Intravenous (IV) vs intrahepatic arterial (IHA) 5-FU/leucovorin for colorectal (CRC) liver metastasis: preliminary results of the MRC CRO5/EORTC 40972 randomised trial. [Abstract] Eur J Cancer 37 (suppl 6): A-955, s257, 2001.